CLINICAL TRIAL: NCT07323238
Title: Hong Kong Cardiogenic Shock Initiative
Acronym: HK CSI
Status: Not yet recruiting | Type: Observational
Sponsor: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Collaborators: Queen Elizabeth Hospital, Hong Kong (Other); Tuen Mun Hospital, Hospital Authority, Hong Koong (Unknown)
Responsible Party: Principal Investigator, Dr So Chak Yu kent, Clinical Asisstant Professor, Prince of Wales Hospital, Shatin, Hong Kong
Other Study IDs: 2025.671
Record Dates: First submitted 2025-12-03; First posted 2026-01-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Cardiogenic Shock Acute; STEMI - ST Elevation Myocardial Infarction; Cardiogenic Shock; Cardiogenic Shock Post Myocardial Infarction; Mechanical Circulatory Support
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GSCI-eligible: Cases that need mechanical cardiovascular support and meet all GSCI incluision and exclusion criterias
- GSCI-ineligible: All other cases with Cardiogenic shock but do not meet all GSCI incluision and exclusion criterias

SUMMARY:
Acute myocardial infarction complicated by cardiogenic shock (AMI-CS) is a severe condition with high mortality. Early revascularization and Impella device (Abiomed) support improve outcomes. Observational studies like the National Cardiogenic Shock Initiative (NCSI), Inova-Shock registry, and J-PVAD (Japan registry for percutaneous ventricular assist device) registry emphasize the importance of structured care systems when using mechanical circulatory support (MCS).

Following the release of the Danger Shock trial, MCS use is expected to rise. Hospitals will need to monitor practices and work with payers to ensure coverage. Using regional real-world data can assist this process, making the collection and analysis of MCS outcomes essential.

The NCSI (NCT03677180) aimed to evaluate outcomes with a protocolized approach prioritizing rapid diagnosis, timely MCS delivery, and invasive hemodynamic monitoring via pulmonary artery (PA) catheters. The study involved 406 patients from 2016 to 2020, with an average age of 64 years. Most (67%) had shock, with 85% on vasoactive drugs. Witnessed outof-hospital cardiac arrest occurred in 17%, and in-hospital arrest in 30%. During MCS implantation, 9% were actively resuscitating. Patients mostly in SCAI stage C/D (73%) and stage E (27%) presented with low blood pressure, high lactate, and reduced cardiac power output. About 70% received MCS before PCI, with 90% using PA catheters. Most had STEMI, with median door-to-support and door-to-balloon times of about 78 and 81 minutes. Survival rates were high: 99% procedural, 79% to discharge, 77% at 30 days, and 62% at one year for stage C/D shock. Patients with stage E shock had lower survival. Early use of MCS improved hemodynamics and survival. Further research, like the CERAMICS (Can Escalation Reduce Acute Myocardial Infarction in Cardiogenic Shock) study, aims to refine escalation strategies. The Danger Shock trial highlighted the importance of minimizing complications such as bleeding, limb ischemia, haemolysis, and kidney injury.

Currently in Hong Kong, prevalence of CS among AMI patients is 5-10%, in-line with global statistics. Among which, 30-day and 1-year mortality of AMI-CS patients in Hong Kong was reported at 29% and 39.5% respectively. Although the use of MCS has been shown in the above overseas studies to improved survival rates of AMI-CS patients, the utilisation rate of MCS among AMI-CS patients in Hong Kong was reported at 36.5% in a previous single-centre study, limited by an array of factors including limited device availability, allocations of resources and patient selection strategy, lack of region-specific evidence and device affordability. Global Cardiogenic Shock Initiative (GCSI) is an ongoing international multicenter registry involving centers from USA, Germany, and Hong Kong, and focus on the outcomes of AMI-CS patients received Impella support. The GCSI is expanding to many other regions. In the Hong Kong Cardiogenic Shock Initiative (HK-CGSI) study we aim to include sites with experience in MCS, all of whom have the capability of MCS escalation and evaluate outcomes across these centers.

The goal is not only to capture the effects of previously established best practices but gain insights into regional best practices, and together with data from the global cardiogenic shock initiative (GCSI), to better establish the adoption of novel best practices and their effect on complication rates.

In parallel to GCSI-eligible cohort, i.e. Impella used as the first supporting device for patients with AMI-CS, given the significant portion of patients who could not receive MCS under current limitations in Hong Kong, in the HK-CSI, we will include also the GCSI-ineligible cohort, i.e. AMI-CSI without using Impella or not as the first MCS used, to understand the full picture of clinical outcomes of AMI-CS patients of Hong Kong.

The HK-CSI study is an observational registry solely and not a treatment study. This single-arm registry captures data generated during procedures which are considered standard of care. Participation in this registry will be performed with waiver of consent of the patient and will have no influence on the type and extent of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myocardial infarction (AMI) with the ECG and/or biomarker evidence of S-T elevation myocardial infarction (STEMI) or non -S-T elevation myocardial infarction (NSTEMI)
* Cardiogenic Shock is defined as presence of at least two of the following

  1. Hypotension (systolic blood pressure ≤ 100 mmHg, or inotropes/vasopressors to maintain systolic blood pressure ≥ 100 mmHg)
  2. Evidence of end organ perfusion: elevated serum lactate levels (venous or arterial), cool extremities, oliguria/anuria
  3. Hemodynamic criteria represented by cardiac index of <2.2 L/min/m² or a cardiac ≤ 0.6 watts
* Patient is supported with a transvalvular MCS as the initial device (criteria for GCSI-eligible Cohort)
* Patients undergo PCI within 12 hours of hospital presentation (criteria for GCSI-eligible Cohort)
* Subject or legally designated representative (LDR) has provided written informed consent. For patients not able to provide consent, data collection will be conducted in retrospective manner with study consent waived.

Exclusion Criteria:

* Unwitnessed out of hospital cardiac arrest or any cardiac arrest in which return of spontaneous circulation (ROSC) is not achieved within 20 minutes
* Patients demonstrate any signs of anoxic brain injury prior to the INDEX PCI (signs of anoxic injury include, posturing, seizures).
* IABP placed prior to MCS (criteria for GCSI-eligible Cohort)
* Septic, anaphylactic, hemorrhagic, and neurologic causes of shock
* Non-ischemic causes of shock/hypotension (pulmonary embolism, pneumothorax, myocarditis, tamponade, etc.)
* Active bleeding for which MCS in contraindicated
* Recent major surgery for which MCS is contraindicated
* Mechanical complication of AMI (acute ventricular septal defect (VSD) or acute papillary muscle rupture)
* Known left ventricular thrombus for which MCS in contraindicated (criteria for GCSI-eligible Cohort)
* Mechanical aortic prosthetic valve (criteria for GCSI-eligible Cohort)
* Contraindication to intravenous systemic anticoagulation which precludes placement of MCS.

Patients who fulfills all Eligibility Criteria would be recruited and considered GSCI-eligible. AMI-CS patients that did not use MCS, ie. Not fulfiliing both Inclusion Criteria 3, 4, would not be considered screen failure and would still be screened and recruited into HKCSI GCSI-ineligible cohort. Likewise, patients who meet any of Exclusion Criteria will not be GCSI-eligible. Specifically, patients who met exclusion criteria 3, 9, 10 only will be recruited into GCSI-ineligible cohort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HKCSI will approximately include 320 cases over 5 years. For subjects in GCSI-eligible cohort (expect n=80), data will be shared with GCSI Study Team and performed together with their Global Database. Analysis of the whole HKCSI cohort will be conducted locally. Study sites will screen all acute myocardial infarction complicated by cardiogenic shock patients, NSTEMI and STEMI, for participation in this trial.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-04-01 (Estimated); Study Completion 2030-10-02 (Estimated)

PRIMARY OUTCOMES:
MCS escalation rate during index hospitalisation | Perioperative
  MCS escalation rate of AMI-CS patient with use of MCS
1-year mortality | 1-year
  1-year mortality of AMI-CS patient with use of MCS
1-year mortality | 1-year
  1-year mortality of AMI-CS patient without use of MCS
30-day mortality | 30-day
  30-day mortality of AMI-CS patient without use of MCS
30-day mortality | 30-day
  30-day mortality of AMI-CS patient with use of MCS

SECONDARY OUTCOMES:
180-day Mortality rate | 180-day
  180-day mortality rate of AMI-CS patient with use of MCS
180-day Mortality rate | 180-day
  180-day mortality rate of AMI-CS patient without use of MCS
30-day MCS escalation rate | 30-day
  MCS escalation rate of AMI-CS patient with use of MCS at 30-day
180-day MCS escalation rate | 180-day
  MCS escalation rate of AMI-CS patient with use of MCS at 30-day
360-day MCS escalation rate | 360-day
  MCS escalation rate of AMI-CS patient with use of MCS at 30-day
Rate of In-Hospital Access Site Bleeding | Perioperative
  Rate of In-Hospital Access Site Bleeding rated by BARC Bleeding Events during index hospitalization
Rate of acute kidney injury | Perioperative
  Acute kidney injury (AKI) per KIDIGO (modified AKIN level >=2) during index hospitalization
Rate of Acute Limb Ischemia | Perioperative
  Acute Limb Ischemia requiring fasciotomy and/or amputation during index hospitalization
Lactate level | Perioperative
  Lactate Clearance during index hospitalization
Blood Transfusion rate | Perioperative
  Rate of Blood Transfusion due to Consumption during index hospitalization
Blood Transfusion rate | Perioperative
  Rate of Blood Transfusion due to Hemolysis during index hospitalization
MCS escalation rate | Perioperative
  MCS escalation rate of AMI-CS patient with use of MCS During index hospitalisation
MCS escalation rate | First 12 hours during index hospitalisation
  MCS escalation rate of AMI-CS patient with use of MCS During index hospitalisation within 12 hours of hemodynamic findings
Rate of MCS re-introduction after removal | Perioperative until discharge
  Rate of MCS re-introduction after removal in AMI-CS patient with use of MCS
Access Site Complication rate | within 48 hours of MCS removal
  Rate of MCS Access Site Complications within 48 hours of MCS removal
Access Site bleeding rate | within 48 hours of MCS removal
  Rate of MCS Access Site bleeding within 48 hours of MCS removal

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No